CLINICAL TRIAL: NCT06624384
Title: Efficacy and Safety of Topical Cyclosporine 0.05% (Restasis) and Lifitgrast (Xiidra) on the Ocular Surface Symptom After Photorefractive Keratectomy (PRK) in Feiz Hospital, Isfahan, 2024
Brief Title: Efficacy and Safety of Topical Cyclosporine 0.05% and Lifitgrast on the Ocular Surface Symptom After Photorefractive Keratectomy in Feiz Hospital, Isfahan, 2024
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mohsen Pourazizi (Other)
Responsible Party: Sponsor-Investigator, Mohsen Pourazizi, Assistant Professor of Ophthalmology, Isfahan University of Medical Sciences
Organization: Isfahan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IR.MUI.MED.REC.1403.129
Record Dates: First submitted 2024-09-24; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Ocular Surface Symptom; Ocular Surface Disease; Eye Pain; Eye Inflammation
Keywords: PRK- ocular surface symptom - cyclosporine 0.05% - Lifitgrast (Xiidra)
MeSH Terms: conditions — Eye Pain; Endophthalmitis | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Group 1: Drug group (topical cyclosporine 0.05% and Lifitgrast) (Active Comparator): Group 1: In this group, cyclosporine 0.05% drops are poured into one eye and Lifitgrast drops are poured into the opposite eye.
  Interventions: Drug: Group 1 drug
- Group 2: drug and placebo (cyclosporine 0.05%-Artlac) (Active Comparator): Group 2: In this group, cyclosporine 0.05% drops are poured into one eye and artelac drops are poured into the opposite eye.
  Interventions: Drug: Group 2: Drug and placebo
- Group 3: drug and placebo (Lifitgrast-Artlac) (Active Comparator): Group 3: In this group, Lifitgrast drops are poured into one eye and artelac drops are poured into the opposite eye.
  Interventions: Drug: Group 3: Drug and palcebo

INTERVENTIONS:
Drug: Group 1 drug — Group 1: In this group, the aim is to compare 2 drugs, cyclosporine 0.05% and Lifitgrast . In one eye, cyclosporine 0.05% eye drops are randomly poured and in the opposite eye, Lifitgrast eye drops are poured.
  Other Names: drug
  Arms: Group 1: Drug group (topical cyclosporine 0.05% and Lifitgrast)
Drug: Group 2: Drug and placebo — Group 2: In this group, the aim is to compare 2 drugs, cyclosporine 0.05% and Artelac artificial tear as a placebo. In one eye, cyclosporine 0.05% eye drops are randomly poured, and in the opposite eye, Artelac artificial tear are poured.
  Arms: Group 2: drug and placebo (cyclosporine 0.05%-Artlac)
Drug: Group 3: Drug and palcebo — Group 3: In this group, the aim is to compare 2 drugs, Lifitgrast and Artelac artificial tear as a placebo. In one eye, Lifitgrast eye drops are randomly poured, and in the opposite eye, Artelac artificial tear are poured.
  Arms: Group 3: drug and placebo (Lifitgrast-Artlac)

SUMMARY:
The goal of this clinical trial is to compare the administration of 2 drugs, cyclosporine 0.05% (Restasis) and Lifitgrast (Xiidra) before PRK, in reducing the ocular surface symptom of patients after PRK. The main questions it aims to answer are:

1- Does the use of cyclosporine 0.05% (Restasis) and Lifitgrast (Xiidra) before photorefractive keratectomy surgery (PRK) reduce ocular surface symptom such as eye pain, redness, and inflammation in conjunctivitis in patients? Researchers will compare cyclosporine 0.05% (Restasis) and Lifitgrast (Xiidra) to a placebo (Artelac artificial tears) to see if cyclosporine 0.05% and Lifitgrast works to reduce ocular surface symptom.

Participants will:

Take drug cyclosporine 0.05% and Lifitgrast or a Artelac 30 minutes before surgery Visit the clinic 6 hours, one day, three days and one week after photorefractive keratectomy (PRK) for checkups and tests

DETAILED DESCRIPTION:
Considering the increasing importance of reducing eye symptoms of patients after PRK surgery and the impact of this issue on the quality of life of patients, as well as the lack of sufficient studies on the effect of different drugs in this field and comparing their effects, which ultimately lead to the decision and clinical application of this Regarding the category of drugs, the present study aims to compare the administration of 2 drugs, cyclosporine 0.05% and Lifitgrast before PRK, in reducing the eye symptoms of patients after PRK.

In this study, 15 minutes before the start of photorefractive keratectomy surgery, we divide the patients into 3 random groups and according to the following plan, we put the drops into the eyes of the patients.

The first group: one eye drop cyclosporine 0.05% - opposite eye drop Lifitgrast The second group: one eye with 0.05% cyclosporine drops - the opposite eye with Artlac artificial tear drops The third group: one eye with Liffitgrast drops - the opposite eye with Artlac artificial tear drops Patients will be evaluated and examined according to variables 6 hours, one day, three days and one week after the operation. To check the symptoms of patients from standard questionnaires including Ocular surface disease index (OSDI), visual analogue scale (VAS) Wong-Baker FACES, Efron is used.

ELIGIBILITY:
Inclusion Criteria:

Age above 18 years Myopia and myopic astigmatism The stability of the patients refraction over the past year Not using contact lenses at least 3 weeks before the operation Absence of history of KCN and any type of corneal ectasia in the patient himself or his first degree family No history of previous eye surgery and eye trauma Absence of active eye diseases, corneal dystrophy, retinal diseases, glaucoma, dry eyes of any degree.

Absence of systemic diseases that can potentially disrupt wound healing, including diabetes, vascular collagen diseases, and pregnancy.

Not taking inhaled or systemic steroids actively or within 3 months before the procedure Absence of anisometropia Not using any systemic and topical analgesia during the last week

Exclusion Criteria:

The patients lack of consent to continue the study Failure to visit the patient for follow-up The occurrence of any complications during the patients surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
average eye inflammatory symptoms in eyes treated with cyclosporine 0.05%, Lifitgrast and Artlac 6 hours, one day, three days and one week after photorefractive keratectomy. | 1 week
  The average inflammatory symptoms of the ocular surface symptoms including pain, burning and itching, redness and conjunctivitis in eyes treated with cyclosporine 0.05%, Lifitgrast and Artlac 6 hours, one day, three days and one week after photorefractive keratectomy(PRK) using a standard questionnaire including Ocular Surface Disease Index (OSDI), Visual Analogue Scale (VAS), Wang Baker FACES and Efron is measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Isfahan University of Medical Sciences, Feiz Hospital, Isfahan, Isfahan, Isfahan, Iran